CLINICAL TRIAL: NCT02711644
Title: Promoting Healthy Weights, Lifestyles and Nutrition During Pregnancy Through Innovative Counselling Methods
Brief Title: Promoting Healthy Weights, Lifestyles and Nutrition in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Danone Institute International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00054360
Record Dates: First submitted 2015-12-22; First posted 2016-03-17 (Estimated); Last update posted 2022-07-19 (Actual); Status verified 2016-09

CONDITIONS: Pregnancy
Keywords: Pregnancy; Prenatal; Nutrition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supportive Lifestyle Counselling (Experimental): Two supportive lifestyle counselling sessions with Registered Dietitian from study entry to 34 weeks.gestation.
  Interventions: Behavioral: Supportive Lifestyle Counselling; Behavioral: Standard Lifestyle Counselling
- Standard Lifestyle Counselling (Active Comparator): Two standard counselling sessions with Registered Dietitian from study entry to 34 weeks gestation
  Interventions: Behavioral: Standard Lifestyle Counselling

INTERVENTIONS:
Behavioral: Supportive Lifestyle Counselling — Each participant will meet with the intervention Registered Dietitian twice in pregnancy and have two follow-up phone calls. Participants in this group will have on-going, supportive discussions with the intervention Registered Dietitian about healthy lifestyles in pregnancy. Discussion topics with the intervention Registered Dietitian at each visit will be participant-centered, allowing the participant to guide the conversation. These conversations will be reinforced at every future contact made throughout pregnancy.
  Arms: Supportive Lifestyle Counselling
Behavioral: Standard Lifestyle Counselling — Each participant will meet in person with their respective Registered Dietitian twice in pregnancy and have two follow-up phone calls. At these visits, each participant will complete questionnaires and have anthropometric assessments (height/weight). From home, each participant will also complete online questionnaires at week 26, and week 34. Postpartum,each participant will complete an online questionnaire. Optional postpartum participation includes a focus group in the postpartum period and the option to meet with a Registered Dietitian postpartum.

SUMMARY:
Research has shown that a woman's lifestyle during pregnancy can predict the future health of a mother and her child. Improving the health of a mother during pregnancy can lead to the best health outcomes for mother and child in the short and long-term period. Currently there is a lack of understanding about how best to support women to achieve healthy weights during pregnancy. The aim of this study is to understand if additional lifestyle support, such as discussions about healthy eating and physical activity provided by a healthcare provider throughout pregnancy can help women achieve weights concordant with gestational recommendations.

The healthcare providers in this study will be Registered Dietitians (RD). The intervention RD will be trained in Healthy Conversations, a supportive method of communication that utilizes open-ended questions to support patient-centered behaviour change. This allows women to explore health issues, identify barriers and discover solutions for improving their own health. This supportive prenatal counselling will occur with the intervention group concurrently while completing lifestyle questionnaires with the study RD. During these conversations, health goals will be made and will be followed up at future visits. The control group will complete the lifestyle questionnaires with the control RD; they will not receive additional lifestyle support at these visits. Women will be randomized into one of the two study groups and will be blinded to their study allocation. All participants will complete two in person visits and two follow-up telephone calls. Data will be collected on diet, physical activity, gestational weight gain, delivery, and infant outcomes.

After this research is complete, the investigators hope to better understand the quantity and quality of additional support that may help women in Alberta achieve guideline concordant weight gain during pregnancy. If interventions can help women gain weight within the guidelines, pregnancy-related complications can be reduced. This information is also aimed at providing a better understanding of healthcare system requirements (i.e., type of providers and care model) in supporting women achieve healthy weights in pregnancy. The findings from this project have the potential to improve prenatal healthcare delivery across the province.

DETAILED DESCRIPTION:
Study Objectives:

1. To examine the efficacy of a supportive prenatal counselling (intervention) vs. standard prenatal care (control) in promoting appropriate weight gain and dietary intake among pregnant women.
2. To describe pregnant women's and the RD's perceptions of the strengths, limitations, effectiveness and satisfaction with the supportive prenatal counselling (intervention) vs. standard care (control).

Study Design:

Seventy women < 20 weeks gestation will be recruited to participate in this randomized control trial. Interested women will be screened in person or by telephone by research staff to determine eligibility. During screening, participants will provide their self-reported height and pre-pregnancy weight. After eligibility is determined, the eligible participants will be stratified by pre-pregnancy body mass index (BMI). Block randomization will occur within each stratum to determine group assignment. Participants will be blinded to their group assignment, as all participants will follow the same study timeline and the visits will consist of the same procedures (completing questionnaires, measuring anthropometrics). During the visit, the control group will take part in routine prenatal care conversations with a Control RD, while the intervention group will receive conversations framed in a Healthy Conversations and 5As approach with the (different) RD. This is deemed as supportive prenatal counselling in our study. The investigators do not anticipate the participants would know the difference. At time of screening, the Baseline Visit will be scheduled with the respective RD. One RD will be responsible for participant contact and data collection from each group. Baseline and follow up appointments will take place at the Clinical Research Unit (CRU)/Human Nutrition Research Unit (HNRU), 2nd floor of the Li Ka Shing Centre for Health Research Innovation. All questionnaires used in this study will be online and available either in RedCap or through ASA24-CANADA-2014 (a specific dietary recall system). All participants will continue to receive prenatal care through their normal care providers, usually a Family Physician and/or Obstetrician/Gynecologist.

At the baseline visit, study staff will confirm participant eligibility, answer any questions, and review the "Information & Consent Form". Women will be asked to provide their healthcare number and permission to collect information from the Antenatal and Delivery and Birth records. For each group, the respective RD will guide participants in completing: the "Baseline Lifestyle Questionnaire" and a ASA24-Hr dietary recall. Each participant's weight and height will be measured. All participants will be provided with a package of general printed resources that contain relevant health information for pregnancy. After each visit and phone call, the RDs will record notes in the participant's study chart. At 28 and 34 weeks gestation, the respective RDs will call the participants to remind them to complete the dietary recalls and/or book the next clinic visit. For the intervention group, the RD will follow-up with goals previously set (if any). At approximately 30 weeks gestation, study visit 2 will occur to complete the "30 Week Lifestyle Questionnaire" for both the intervention and control groups. At 34 weeks, all participants will be sent the link in their email to complete the "34 Week Lifestyle Questionnaire" and the ASA-24 Hr recall. At approximately 4-6 weeks postpartum, all participants will receive a link to the "Postpartum Questionnaire". Participants in both groups will be asked if they would like to take part in a post-study focus group to discuss their perceptions of the strengths, limitations, effectiveness and satisfaction with the study. A separate focus group will be conducted for each arm of the study and will be facilitated by study staff that is not known to the participants. Participants who would like to meet with a RD for postpartum nutrition counselling will have the opportunity to schedule a session; no data collection will occur at this point.

For the intervention group (n=35), the process of completing the questionnaires and assessments will be framed using a Healthy Conversation approach. This includes the use of open-ended questions that enable participant-centered discussions on topics related to healthy weights, healthy eating, and other lifestyle factors in pregnancy. Discussion topics will be participant-centered, allowing the participant to guide the conversation. This type of exploratory counselling allows the participant to understand barriers they face and come up with solutions that will work within their life. These conversations will be reinforced at each in-person session and during each telephone follow-up. The intervention group can contact the study RD and ask questions via phone, email, video call and/or text message throughout pregnancy. The study team will record the quality and the quantity of all contacts with each participant.

For the control group (n=35), the RD will help participants complete the questionnaires and assessments (data collection only) without discussion of specific pregnancy-related topics. Questions directed at the RD will be answered within the scope of the RD's practice; however, not additional supportive prenatal counselling will be provided at these study visits. Participants in the control group will not receive any further follow-up other than the 2 study visits and 2 phone calls.

The investigators will also collect data from the 2 RDs throughout this study. The intervention RD will complete notes after each contact with participants. The mode of contact, total minutes, topic of discussion, goals made and amount of minutes a Healthy Conversation was held with the participants, will be noted. The RDs will ask a random sample of participants in each arm for permission to audio-record some of their visits to examine the fidelity and competency of the RD in delivering the intervention using Healthy Conversation Skills. Both RDs will record their perceptions of the strengths, limitations, and satisfaction with the study arm they administer to evaluate both protocols through their visit notes. Additionally, at the end of the study, the RDs will each complete a study reflection. These notes will be qualitatively analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 20 years of age
* Between 8-20 weeks gestation
* Singleton pregnancy
* Can read and speak English
* Has Internet and telephone access
* Can make the Baseline visit by 24 weeks gestation
* Willingness to provide pre-pregnancy weight and height
* Willingness to provide Alberta Healthcare Number (PHN)
* Willingness to be randomized
* Will be blinded to group allocation.

Exclusion Criteria:

* Smoker
* Incompetent cervix (previous or present diagnosis)
* Complete/total placenta previa
* Type I, Type II, Gestational Diabetes
* Hypothyroidism (low thyroid function)
* Hyperthyroidism (overactive thyroid)
* Present eating disorder
* Pregnancy-Induced Hypertension (PIH) with adverse features (ie: edema)
* Physical activity is contraindicated
* Currently receiving counselling from a Dietitian
* Currently participating in another lifestyle program
* Receiving prenatal care from a Midwife

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2015-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Weight change from pre-pregnancy to end of pregnancy | pre-pregnancy, study entry (8-24 weeks gestation), gestational week 30, delivery
  difference between self-reported pre-pregnancy weight and highest weight in pregnancy

SECONDARY OUTCOMES:
Type of Labour | Delivery
  from prenatal/delivery record
Mother's perceptions of quality of prenatal care | 1 month Postpartum
  Quality of prenatal care Questionnaire (Sword, Heaman 2013)
Rate of weight gain | From pre-pregnancy through delivery
  calculated from weights recorded on prenatal record
Pregnancy Physical Activity Questionnaire (PPAQ) | Baseline, week 30 and week 34 gestation
  A calculation is provided by the investigators whom created the PPAQ. Each activity is multiplied by an intensity to provide an average weekly energy expenditure.
Changes in dietary quality | Baseline, week 30 and week 34 gestation
  Food and nutrient intake determined by 24 hour dietary recall
Augmentation used during delivery | Delivery
  from prenatal/delivery record (administration of oxytocin - yes/no)
Type of Birth | Delivery
  from prenatal/delivery record
Degree of Perineal Tearing | Delivery
  from prenatal/delivery record (degree of Perineal Tearing - nil, 1, 2, 3)
Blood loss | Delivery
  from prenatal/delivery record
Duration of Labour | Delivery
  from prenatal/delivery record
Cord pH | Delivery
  from prenatal/delivery record
Meconium Fluid | Delivery
  from prenatal/delivery record
Breastfeeding initiation in hospital | Delivery
  from Delivery Record
NICU Admission | Delivery
  from Delivery Record
Infant sex | Delivery
  from Delivery Record
Gestational age at birth | Delivery
  from Delivery Record
Infant birth weight | Delivery
  from Delivery Record
Infant birth weight percentile | Delivery
  from Delivery Record
Infant birth length | Delivery
  from Delivery Record
Infant birth length percentile | Delivery
  from Delivery Record
APGAR Score | Delivery
  from Delivery Record

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda Bell, PhD, Principal Investigator — University of Alberta; Donna Manca, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adam LM, Manca DP, Bell RC. Can Facebook Be Used for Research? Experiences Using Facebook to Recruit Pregnant Women for a Randomized Controlled Trial. J Med Internet Res. 2016 Sep 21;18(9):e250. doi: 10.2196/jmir.6404. PMID 27655184
- See also: Study Website — https://enrich.ales.ualberta.ca/Current-Opportunities